CLINICAL TRIAL: NCT06304038
Title: Cost-consequence Analysis of Influenza Vaccination Among the Staff of a Large Teaching Hospital in Rome, Italy: A Pilot Study
Brief Title: Cost-consequence Analysis of Influenza Vaccination in a Teaching Hospital in Rome
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Laurenti Patrizia, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2018
Record Dates: First submitted 2023-03-11; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Influenza Vaccine; Cost-Benefit Analysis
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccinated subjects: Healthcare workers that received quadrivalent split inactivated non-adjuvanted flu vaccine Fluarix Tetra in a single administration
  Interventions: Drug: Flu Vaccine
- Unvaccinated subjects: Healthcare workers that did not received flu vaccine

INTERVENTIONS:
Drug: Flu Vaccine — Administration of quadrivalent split inactivated non-adjuvanted flu vaccine Fluarix Tetra
  Groups: Vaccinated subjects

SUMMARY:
Flu vaccination, as well as being effective to prevent seasonal influenza, decreases staff illness and absenteeism and reduces costs resulting from loss of productivity. Despite the effectiveness of flu vaccination, the seasonal coverage among healthcare workers is usually low. The aim of this retrospective observational study is to analyze the vaccination coverage rate among all employees (healthcare workers and administrative staff) of a large teaching hospital in Rome during the 2017-2018 influenza season, to perform a cost-consequence analysis of influenza vaccination (by evaluating the absenteeism due to illness in the epidemic period), and to assess the impact of vaccination in terms of both costs and sick days.

ELIGIBILITY:
Inclusion Criteria:

• Healthcare workers at Fondazione Policlinico Universitario "A.Gemelli" IRCCS

Exclusion Criteria:

• Healthcare workers not working at Fondazione Policlinico Universitario "A.Gemelli" IRCCS

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is represented by all employed healthcare workers of the FPG amounting to approximately 5000 (data provided by the Human Resources Department of the Hospital in December 2017).
  The case group consists of all healthcare workers vaccinated in the 2017-2018 season at the specially designated facilities within the Teaching Hospital, filed on special registers.
  The control group consists of healthcare workers who were not vaccinated in the 2017-2018 season at the specially designated facilities within the Teaching Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5483 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-04-29 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the quadrivalent vaccine | 33 weeks
  Effectiveness of the quadrivalent vaccine in reducing the number of working days lost due to influenza syndrome
Economic impact of the quadrivalent vaccine | 33 weeks
  Economic impact (for the company and society) of vaccination as part of a vaccination campaign on the healthcare workers of the teaching hospital.

SECONDARY OUTCOMES:
Expected economic savings for each one percentage point increase in vaccination coverage | 33 weeks
  Expected economic savings for each one percentage point increase in coverage on the health personnel of the teaching hospital
Non-economic incentives for healthcare personnel who decide to vaccinate | 33 weeks
  Non-economic incentives for healthcare personnel who decide to vaccinate, in view of the financial savings for the company, linked to increased vaccination coverage

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "A.Gemelli" IRCCS, Rome, Italy